CLINICAL TRIAL: NCT03966599
Title: Comparison of Hemodynamic Stability and Pain Control Between Two Anesthesia Positions of Lateral and Prone in Patients Undergoing Percutaneous Nephrolithotomy; a Randomized Controlled Trial Study
Brief Title: Comparison of Hemodynamic Stability and Pain Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Hamidreza Shemshaki, Director, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 121333P
Record Dates: First submitted 2019-05-17; First posted 2019-05-29 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Percutaneous Nephrolithotomy
Keywords: Percutaneous Nephrolithotomy; Analgesic; hemodynamic status
MeSH Terms: interventions — Pain Measurement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lateral position (Active Comparator): The patient position was changed to lateral during surgery
  Interventions: Diagnostic Test: Pain; Diagnostic Test: Hemodynamic changes
- prone position (Active Comparator): The patient position was changed to prone during surgery
  Interventions: Diagnostic Test: Pain; Diagnostic Test: Hemodynamic changes

INTERVENTIONS:
Diagnostic Test: Pain — Patient's pain in order to VAS
Diagnostic Test: Hemodynamic changes — changes in hemodynamic states

SUMMARY:
This study was designed to evaluate whether patient position (lateral vs. prone) has affect on the need for analgesia and onset of pain after surgery.

DETAILED DESCRIPTION:
Percutaneous Nephrolithotomy is the preferred surgical treatment in many cases of kidney stones which is performed in different positions such as prone, lateral, and supine. However, we do not have enough evidence comparing prone and lateral positioning regarding the need for analgesia and onset of pain after surgery. This study was designed to evaluate whether patient position (lateral vs. prone) has affect on the need for analgesia and onset of pain after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were age between 18-65 years,
* having kidney stones; consent for spinal anesthesia,
* ASA classes (American Society of Anesthesiologists class) of 1 and 2 (patients without any cardiovascular or respiratory disorders)
* superior and median ureter larger than 20 mm in diameter.

Exclusion Criteria:

* those with coagulation defects,
* severe pain requiring more than one dose of fentanyl,
* considerable rise of blood pressure or heart rate during the operation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2018-01-02 (Actual); Study Completion 2018-02-03 (Actual)

PRIMARY OUTCOMES:
pain intensity in VAS score and need for analgesics in milligram | at one year after surgery
  determining pain with visual analogue scale (VAS) and need for analgesics (milligram) in lateral versus prone position. The visual analogue scale (VAS) is usually presented as a 100-mm horizontal line on which the patient's pain intensity is represented by a point between the extremes of "no pain at all" and "worst pain imaginable." Its simplicity, reliability, and validity, as well as its ratio scale properties, make the VAS the optimal tool for describing pain severity or intensity.

SECONDARY OUTCOMES:
hemodynamic state | at one year after surgery
  changes in blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Hamidreza Shemshaki, MD, Study Director — shahid beheshti university of medical sciences, tehran, iran